CLINICAL TRIAL: NCT04983823
Title: Persistent Cardiovascular Effects of COVID-19 Viral Infection Trial (PERCEIVE): A Randomised Controlled Trial of the Role of Optimal Cardioprotection Strategies to Prevent Heart Failure
Brief Title: Persistent Cardiovascular Effects of COVID-19 Viral Infection Trial (PERCEIVE)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baker Heart and Diabetes Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 28/21
Record Dates: First submitted 2021-07-29; First posted 2021-07-30 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Heart Failure
Keywords: Heart failure; COVID
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Randomization to CC-DMP or usual care
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor will receive study data based on pooled de identified dataset.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Heart failure intervention (Cardiac COVID Disease Management Plan (CC-DMP) (Experimental): 1. Optimization of pharmacotherapy:
     This will be performed by a supervising clinician and will comprise treatment with angiotensin-converting enzyme inhibitor (ACEi, Ramipril) and beta blocker (Metoprolol) for cardioprotection.
  2. Exercise intervention: Individualized training program will be provided by an exercise physiologist
  Interventions: Other: Heart Failure intervention (Cardiac COVID Disease Management Plan (CC-DMP)
- Usual care (Active Comparator): All medical management for participants allocated to this group will be at the discretion of their usual care healthcare professional(s).
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Heart Failure intervention (Cardiac COVID Disease Management Plan (CC-DMP) — A clinical review to ensure optimal risk factor control and cardioprotection along with exercise intervention.
  Arms: Heart failure intervention (Cardiac COVID Disease Management Plan (CC-DMP)
Other: Usual care — This will be provided by participants' usual healthcare professional(s).
  Arms: Usual care

SUMMARY:
This is a prospective study in which a process of identifying and improving a reduction of functional capacity in COVID-19 survivors >50 years old.

The overall goal of this study to identify the feasibility and value of risk-guided medical therapy and exercise intervention in COVID-19 survivors.

DETAILED DESCRIPTION:
Participants enrolled in this study will be randomized to a cardio-COVID disease management plan (CC-DMP) that involves the use of VO2 testing and surveillance imaging to detect reduced functional capacity and subclinical left ventricular dysfunction (LVD), clinical review to ensure optimal risk factor control and cardio-protection and exercise intervention. The program will be delivered over a period of 24 months.

The outcome from this study will show that subclinical LVD is common among COVID-19 survivors, and a CC-DMP is feasible in reducing HF risk factors in this sub group of survivors.

ELIGIBILITY:
Inclusion Criteria:

1. History of COVID-19 infection
2. Live within a geographically accessible area for follow-up

Exclusion Criteria:

1. Valvular stenosis or regurgitation of >moderate severity
2. History of previous heart failure (baseline New York Heart Association (NYHA) classification >2)
3. Inability to acquire interpretable images (identified from baseline echo)
4. Contraindications to beta blockers or angiotensin-converting enzyme inhibitors
5. Oncologic (or other) life expectancy <12 months or any other medical condition (including pregnancy) that results in the belief (deemed by the Chief Investigators) that it is not appropriate for the patient to participate in this trial
6. Already taking both angiotensin converting enzyme inhibitors/ angiotensin receptor blockers and beta blockers, or intolerance (or allergy) to both.
7. Mobility impairment that would impact participants' ability to perform exercise
8. Unable to provide written informed consent to participate in this study

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 820 (Estimated)
Dates: Start 2021-11-18 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in exercise capacity | Over a period of 24 months
  Cardio pulmonary fitness (peak oxygen uptake (VO2 peak)) from baseline to follow up.

SECONDARY OUTCOMES:
New onset heart failure | Over a period of 24 months
  Symptoms and signs of heart failure (Framingham criteria)
Change in maximal isometric grip strength | Over a period of 24 months
  Strength (kg) measured by electronic dynamometer
Change on quality of life | Over a period of 24 months
  Change in score on Health related quality of life: Assessment of quality of life 8 Dimension.
  Minimum value 1, Maximum value 4. Higher values indicate worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas H Marwick, MD,PhD,MPH, Principal Investigator — Baker Heart and Diabetes Institute
Locations (1):
- Baker Heart and Diabetes Institute, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No
Data sharing based available on application to the study PI